CLINICAL TRIAL: NCT03768635
Title: Necrotizing External Otitis : Study in a Regional Bone and Joint Infection
Brief Title: Necrotizing External Otitis : Study in a Regional Bone and Joint Infection Reference Center
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Eugénie MABRUT, Clinical Reseacrh Assistant, Hospices Civils de Lyon
Other Study IDs: 18-284
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Bone and Joint Infection
Keywords: otitis
MeSH Terms: conditions — Otitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Necrotizing external otitis: description of necrotizing external otitis
  Interventions: Other: necrotizing external otitis

INTERVENTIONS:
Other: necrotizing external otitis — description of necrotizing external otitis

SUMMARY:
The malignant external otitis is a rare disease which arises more frequently at the elderly and the diabetics patients. To our knowledge, there are few data and it is not wellc known byclinicians. Nevertheless it exposes to neurological complications potentially serious and crippling.

ELIGIBILITY:
Inclusion Criteria:

* patients having had necrotizing external otitis and managed at the Lyon Bone and joint infection refence Center

Exclusion Criteria:

* none

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients having had necrotizing external otitis and managed at the Lyon Bone and joint infection refence Center between 01/01/2006 and 31/01/2018
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Rate of necrotizing external otitis | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  description of necrotizing external otitis: patients, profile of the bacterium, medical and chirurgical treatment, rate

SECONDARY OUTCOMES:
Rate of Treatment Failure | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin. Analyse of risk factor.
Duration of antibiotics | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  Description of the strategies of antibiotic treatments used (double-agent therapy, monotherapy, duration)

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Ferry, Md, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided